CLINICAL TRIAL: NCT04800354
Title: Brief Nurse-led Mindfulness Based Intervention Among Patients Scheduled for Knee and Hip Replacement Surgery
Brief Title: Brief Nurse-led Mindfulness Based Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Adam Hanley, Assistant Professor, University of Utah
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB_00085446: AM_00040605
Record Dates: First submitted 2021-03-07; First posted 2021-03-16 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2022-01

CONDITIONS: Pain; Osteoarthritis, Knee; Osteoarthritis, Hip
MeSH Terms: conditions — Pain; Osteoarthritis, Knee; Osteoarthritis, Hip

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nurse-led Mindfulness Based Intervention (Experimental)
  Interventions: Behavioral: Nurse-led Mindfulness Based Intervention; Behavioral: Nurse-led Pain Psychoeducation
- Nurse-led Pain Psychoeducation (Active Comparator)
  Interventions: Behavioral: Nurse-led Pain Psychoeducation

INTERVENTIONS:
Behavioral: Nurse-led Mindfulness Based Intervention — Nurses will read patients a brief (1 minute) scripted, introduction to mindfulness and then have them listen to a very brief (1 minute 30 second) guided mindfulness practice validated in our prior research to encourage focused attention on breath and body sensations and open monitoring and acceptance of discursive thoughts, negative emotions, and pain. Finally, patients will be given an audio recording of the mindful pain management technique for use any time they experience intense pain or take pain medication before and after surgery.
  Arms: Nurse-led Mindfulness Based Intervention
Behavioral: Nurse-led Pain Psychoeducation — Nurses will provide psychoeducation about pain along with common pain coping strategies, such as rest, ice, and elevation, for use any time they experience intense pain or take pain medication before and after surgery.

SUMMARY:
This is a single-site, two-arm, parallel-group randomized clinical trial (RCT). The feasibility, acceptability, and clinical effects of the nurse-led, very brief, preoperative mindfulness based intervention for hip and knee replacement patients will be investigated relative to nurse-led preoperative pain psychoeducation.

A secondary sub-analysis will compare two different styles of mindfulness practice (mindfulness of breath vs. mindfulness of pain) relative to preoperative pain psychoeducation.

ELIGIBILITY:
Inclusion Criteria:

* 1) Age ≥18,
* 2) Scheduled to undergo unilateral total knee arthroplasty

Exclusion Criteria:

* 1) Cognitive impairment preventing completion of study procedures.
* 2) Current cancer diagnosis,
* 3) Contralateral knee replaced in the previous 3 months,
* 4) Intent to have contralateral knee replaced or other, additional surgical procedure during the study period,
* 5) Intent to add new pain treatments during the study period (except for what is part of the study),
* 6) Other unstable illness judged by medical staff to interfere with study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 127 (Actual)
Dates: Start 2021-02-22 (Actual); Primary Completion 2021-05-20 (Actual); Study Completion 2022-01-10 (Actual)

PRIMARY OUTCOMES:
Change in Pain Intensity Numeric Rating Scale | baseline and after the 15 minute preoperative nurse visit
  Single Likert scale item ranging from 0-10, with 0 indicating no pain and 10 representing the most intense pain imaginable.

SECONDARY OUTCOMES:
Change in Pain Unpleasantness Numeric Rating Scale | baseline and after the 15 minute preoperative nurse visit
  Single Likert scale item ranging from 0-10, with 0 indicating no pain and 10 representing the most unpleasant pain imaginable.
Change in Pain Medication Desire Numeric Rating Scale | baseline and after the 15 minute preoperative nurse visit
  Single Likert scale item ranging from 0-10, with 0 indicating no desire for pain medication and 10 representing a strong desire for pain medication.
Postoperative Patient Reported Outcomes Measurement Information System (PROMIS) Physical Functioning Item Bank, v2.0 | During the 6 weeks prior to surgery and at the 6-week outpatient follow-up appointment
  The PROMIS physical functioning computer assisted test draws from a bank of 123 items all scored on a 5 point Likert scale.
  T-Score distributions are standardized such that a 50 represents the average (mean) for the US general population, and the standard deviation around that mean is 10 points. A high score better physical functioning.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Utah, Salt Lake City, Utah, United States